CLINICAL TRIAL: NCT01516463
Title: Comparison of Collagenase Santyl® Ointment With Antibiotic Ointment in the Outpatient Care of Minor Partial Thickness Burns
Brief Title: Using Santyl or Bacitracin on Second Degree Burns
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 017-101-09-031
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Burn, Partial Thickness
Keywords: burn; partial thickness burn; second degree burn; minor burn; scar; Santyl; Bacitracin; outpatient burn center; scar appearance; Kansas City; University of Kansas Medical Center; KUMC
MeSH Terms: conditions — Burns; Cicatrix | interventions — Bacitracin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collagenase Santyl (Active Comparator)
  Interventions: Drug: Collagenase Santyl
- Bacitracin (Sham Comparator)
  Interventions: Biological: Bacitracin

INTERVENTIONS:
Drug: Collagenase Santyl — Applied topically (2 mm thickness once daily)
  Arms: Collagenase Santyl
Biological: Bacitracin — Applied topically (2 mm thickness) once daily
  Arms: Bacitracin

SUMMARY:
Subjects who have minor, second degree burns may be enrolled in this study. Subjects will receive either Santyl ointment or bacitracin ointment to apply to the burn until it heals. Bandages will be used to keep the burn covered while it heals. Second degree burns generally leave a scar. Once the burn heals, lotion and an appropriate bandage will be used to try to minimize the appearance of a scar.

The study hypothesis is that burns treated with Santyl will have a better scar appearance than burns treated with bacitracin.

Subjects enrolled in this study will make once a week visits to the University of Kansas Medical Center outpatient burn clinic until the burn heals. The burn will be assessed for healing at these visits. Once healed, visits to the clinic will be every 1-3 months for up to 1 year. At these visits, the appearance of the scar will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information. For subjects not able to provide informed consent (e.g., minors), a parent or legally authorized representative must provide consent. Assent must be provided as required by the IRB.
* Age 2 - 75 yrs, either sex, any race.
* Have one or more acute burns which:
* • are thermal, chemical or electrical in etiology
* • in aggregate cover <10% TBSA
* • are each equal to or less than 72 hrs old
* • are each no more than deep partial thickness (2nd degree)
* • are not visibly infected
* Able to take in oral fluids.
* Able to comply with the requirement for daily dressing changes, or have a caretaker who is able to comply.
* Willing to make all required study visits.

Exclusion Criteria:

* Contraindications or hypersensitivity to the use of the test article or their components (e.g., known hypersensitivity to bacitracin).
* Embedded foreign bodies in the burn wound which cannot be immediately removed.
* The burned tissue includes or is within 1 cm of the eye or genitalia.
* Severe perioral burns.
* Airway involvement or aspiration of hot liquids.
* Suspicion of physical abuse.
* Burn wound requires a skin graft.
* Outpatient management of the burn wound is not appropriate.
* Participation in another investigational clinical study within thirty (30) days of the Screening Visit.
* Current or recent (< 6 months) history of severe, unstable, or uncontrolled neurological, cardiovascular, gastrointestinal, hematological, hepatic, and/or renal disease or evidence of other diseases based upon a review of medical history that, in the opinion of the Investigator, would preclude safe subject participation in the study.
* The Medical Monitor and / or Investigator may declare any subject ineligible for a valid medical reason.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Scar Appearance | 90 Days

SECONDARY OUTCOMES:
Proportion healed at two weeks | 2 weeks after initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint; Dhaval Bhavsar, MD, Principal Investigator — University of Kansas Medical Center